CLINICAL TRIAL: NCT04249128
Title: The Derm Aid Study
Brief Title: Nourishing Hair, Skin & Nails Supplement Study (Derm Aid)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Noho Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2286
Record Dates: First submitted 2020-01-25; First posted 2020-01-30 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Hair Loss; Skin Laxity; Cosmetic Acne; Nails; Soft; Skin Aging
MeSH Terms: conditions — Alopecia; Cutis Laxa | interventions — Keratins; Ceramides; astaxanthine

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of eight arms. The arms include four combinations of dietary supplements for skin, hair & nail health (Keratin, collagen peptides, pro-berry powder, vegan Keratin, and Astaxanthin). Each supplement formation is included in two arms - one arm is paid, the other arm is free.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is done completely online. Supplements are fulfilled at a central fulfillment center. The study sponsor, nor any care provider, or investigator know what formulation a participant receives until the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Veg Collagen & Keratin Free (Hair Skin Nails) (Experimental): Participants will receive a free 3 month supply of Collagen & Keratin for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Vegetarian Collagen; Dietary Supplement: Keratin
- Veg Collagen Extended with Powder Free (Hair Skin Nails) (Experimental): Participants will receive a free 3- month supply of Collagen & Keratin for Hair, Skin & Nail Health extended with a pro-berry powder
  Interventions: Dietary Supplement: Vegetarian Collagen; Dietary Supplement: Keratin
- Veg Collagen & Keratin $$$ (Hair Skin Nails) (Experimental): Participants will receive a paid 3-month supply of Collagen & Keratin for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Vegetarian Collagen; Dietary Supplement: Keratin
- Veg Collagen Extended with Powder $$$ (Hair Skin Nails) (Experimental): Participants will receive a paid 3-month supply of Collagen & Keratin extended with pro-berry powder for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Vegetarian Collagen; Dietary Supplement: Keratin
- Ceramides and Astaxanthin Free (Skin) (Experimental): Participants will receive a free 3-month supply of ceramides and Astaxanthin for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Ceramides; Dietary Supplement: Astaxanthin
- Ceramides and Astaxanthin Extended with Powder Free (Skin) (Experimental): Participants will receive a free 3-month supply of Ceramides and Astaxanthin for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Ceramides; Dietary Supplement: Astaxanthin
- Ceramides and Astaxanthin $$$ (Skin) (Experimental): Participants will receive a paid 3-month supply of Ceramides and Astaxanthin extended with pro-berry powder for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Ceramides; Dietary Supplement: Astaxanthin
- Ceramides and Astaxanthin Extended with Powder $$$ (Skin) (Experimental): Participants will receive a paid 3-month supply of Ceramides and Astaxanthin extended with pro-berry powder for Hair, Skin & Nail Health
  Interventions: Dietary Supplement: Ceramides; Dietary Supplement: Astaxanthin

INTERVENTIONS:
Dietary Supplement: Vegetarian Collagen — Collagen is a protein made up of amino-acids, which are in turn built of carbon, oxygen and hydrogen.
  Arms: Veg Collagen & Keratin $$$ (Hair Skin Nails); Veg Collagen & Keratin Free (Hair Skin Nails); Veg Collagen Extended with Powder $$$ (Hair Skin Nails); Veg Collagen Extended with Powder Free (Hair Skin Nails)
Dietary Supplement: Keratin — Keratin (/ˈkɛrətɪn/) is one of a family of fibrous structural proteins known as scleroproteins. α-Keratin is a type of keratin found in vertebrates. It is the key structural material making up hair, nails, feathers, horns, claws, hooves, calluses, and the outer layer of skin among vertebrates.
  Arms: Veg Collagen & Keratin $$$ (Hair Skin Nails); Veg Collagen & Keratin Free (Hair Skin Nails); Veg Collagen Extended with Powder $$$ (Hair Skin Nails); Veg Collagen Extended with Powder Free (Hair Skin Nails)
Dietary Supplement: Ceramides — Ceramides are a family of waxy lipid molecules. A ceramide is composed of sphingosine and a fatty acid. Ceramides are found in high concentrations within the cell membrane of eukaryotic cells, since they are component lipids that make up sphingomyelin, one of the major lipids in the lipid bilayer.
  Arms: Ceramides and Astaxanthin $$$ (Skin); Ceramides and Astaxanthin Extended with Powder $$$ (Skin); Ceramides and Astaxanthin Extended with Powder Free (Skin); Ceramides and Astaxanthin Free (Skin)
Dietary Supplement: Astaxanthin — is a naturally-occurring carotenoid found in algae, shrimp, lobster, crab and salmon.
  Arms: Ceramides and Astaxanthin $$$ (Skin); Ceramides and Astaxanthin Extended with Powder $$$ (Skin); Ceramides and Astaxanthin Extended with Powder Free (Skin); Ceramides and Astaxanthin Free (Skin)

SUMMARY:
A 90 day eight arm virtual interventional study looking at the impact of various supplement formulations for improves in hair, skin & nail health via self report, and dermatology assessment via remote dermatologist assessment.

DETAILED DESCRIPTION:
This study is being run entirely on the ProofPilot clinical trial platform. Participants enroll online, submit selfies, and are shipped dietary various dietary supplements containing a one or more of Keratin, Astaxanthin, Collagen Peptides and Pro-berry powder in vegan and non-vegan formats. All participants will receive active ingredients but in various fomulations.

Half the participants will receive the formations for free. The other half will pay a discounted amount for the supplements.

ELIGIBILITY:
Inclusion Criteria:

* Continental US
* ability and willingness to take selfies

Exclusion Criteria:

* skin diease
* use of retinoids
* known allergies
* significant facial hair
* medically relevant skin disease

Ages: 26 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Changes in Self-Report Skin, Hair & Nail Health and Satisfaction | Baseline, 30 Day, 60 Day and 90Day
  A custom self-report survey for participants to self-assess their satisfaction on skin, hair and nail status.
Blinded Dermatology Assessment of Facial Skin health | Baseline 45 day and 90 day
  Comparison over timepoints of physician assessment of facial features at rest and smile to the Glogau & customer wrinkle selfie scale
Participant Acceptability | weekly
  Week by week change and overall analysis of custom survey delivered weekly asking participants to self report acceptability and adherence to treatment regiment over prior week.
Paid versus unpaid particpatnt adherence | 30 and 90 Day
  Comparison of arms with the same intervention, but one paid, one not, to assess impact on adherence

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot Online App (https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to make participant data available to other participants.